CLINICAL TRIAL: NCT07289477
Title: A Phase I/III Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of Intracerebral Putamen Transplantation of NouvNeu001 Injection for Multiple System Atrophy
Brief Title: A Phase I/III Clinical Study to Evaluate NouvNeu001 Injection for Multiple System Atrophy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: iRegene Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NouvNeu004-01
Record Dates: First submitted 2025-11-26; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Multiple System Atrophy - Parkinsonian Subtype (MSA-P)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NouvNeu001 (Experimental): During the enrollment phase for the low-dose cohort, 3 participants will be randomized to the experimental arm to receive a single administration of NouvNeu001 Injection.
  Interventions: Biological: Human Dopaminergic Progenitor Cells
- control (No Intervention): During the enrollment phase for the low-dose cohort, 3 participants will be randomized to the control arm, which will not receive NouvNeu001 Injection.

INTERVENTIONS:
Biological: Human Dopaminergic Progenitor Cells — Single injection of Human Dopaminergic Progenitor Cells into the putamen/striatum region of brain.
  Arms: NouvNeu001

SUMMARY:
This clinical trial is designed to evaluate the safety, tolerability and preliminary efficacy of a single injection of NouvNeu001 (Human Dopaminergic Progenitor Cells Injection) in patients with Multiple System Atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 30 and 70 years (inclusive), regardless of gender.
* The subject understands and agrees to comply with the study procedures and voluntarily provides written informed consent.
* Diagnosed with pathologically confirmed, clinically established, or clinically probable Multiple System Atrophy (MSA) according to the 2022 MDS diagnostic criteria.
* Current treatments for core MSA symptoms are inadequately controlled.
* The duration of MSA-related motor symptoms (parkinsonism and/or cerebellar ataxia) is no more than 5 years.
* Ability to walk without human assistance, defined as being able to take at least 10 steps; the use of assistive devices (e.g., a walker or cane) is permitted.
* Life expectancy of at least 3 years.
* The subject agrees not to participate in any other clinical studies for 24 months following the investigational product administration.

Exclusion Criteria:

* Neurological diseases/disorders other than Multiple System Atrophy, such as Parkinson's disease, Dementia with Lewy Bodies, Essential Tremor, Progressive Supranuclear Palsy, Spinocerebellar Ataxia, Hereditary Spastic Paraplegia, Corticobasal Degeneration, Vascular Parkinsonism, Normal Pressure Hydrocephalus, or Drug-induced/Postencephalitic Parkinsonism.
* Diagnosis of dementia.
* Previous or current receipt of other disease-modifying therapies, or participation in clinical trials of other new drugs or novel therapies.
* Use of medications within the past 3 months that may affect Parkinsonian symptoms, autonomic function, or the evaluation of safety.
* Presence of clinically significant or unstable medical or surgical conditions that may preclude the safe completion of the treatment or confound the treatment outcomes.
* History of or undergoing treatment for recurrent stroke.
* Screening brain MRI shows other significant pathological findings, including but not limited to: cerebral hemorrhage, acute cerebral infarction, aneurysm, vascular malformation, infectious lesions, brain tumors, or other space-occupying lesions (meningiomas or arachnoid cysts with a maximum diameter of less than 1 cm do not warrant exclusion).
* Subjects meeting any of the following criteria indicating advanced disease:

Speech impairment defined by a score of ≥3 on UMSARS Item 1. Swallowing impairment defined by a score of ≥3 on UMSARS Item 2. Walking impairment defined by a score of ≥3 on UMSARS Item 7. Occurrence of falls more than once per week, defined by a score of ≥3 on UMSARS Item 8.

* History of current substance abuse and/or alcohol abuse (within 12 months prior to screening).
* Known allergy to the investigational product(s); or history of allergy to antibiotics or other drugs.
* Positive screening results for active viral infection, including Human Immunodeficiency Virus (HIV), Hepatitis B Surface Antigen (HBsAg), Hepatitis B Core Antibodies, or Hepatitis C Virus (HCV).
* Severe hepatic insufficiency, renal insufficiency, or severe cardiac insufficiency:

Severe hepatic insufficiency: ALT ≥ 2.0 × upper limit of normal (ULN) or AST ≥ 2.0 × ULN.

Severe renal insufficiency: Serum creatinine ≥ 1.5 × ULN or estimated Glomerular Filtration Rate (eGFR) < 40 mL/min/1.73 m².

Severe cardiac insufficiency: New York Heart Association (NYHA) Class 3 or 4.

* History of thrombocytopenia within the past three months, other bleeding disorders, or current receipt of anticoagulant therapy (excluding aspirin at a dose ≤ 100 mg per day).
* Pregnancy, lactation, or planning pregnancy.
* History of Bipolar Disorder, Major Depressive Disorder, Schizophrenia, or other psychotic disorders.
* Subjects judged by the investigator to have suicidal ideation at screening, or a suicide attempt within 6 months prior to screening.
* Contraindications for surgery (e.g., implantation of cochlear implants, pacemakers, defibrillators, history of stereotactic ablation, previous implantation of unilateral/bilateral similar products) or history of other surgeries within the past 6 months deemed by the investigator to potentially affect this trial, or other neurosurgical contraindications.
* Clinically significant cardiac disease defined as: myocardial infarction, NYHA Class III or IV heart failure, uncontrolled coronary spasm, severe uncontrolled ventricular arrhythmia, or evidence of acute ischemia or abnormal conduction system on ECG within 6 months prior to enrollment.
* Diagnosis of malignancy.
* Family history of congenital or inherited immunodeficiency disorders.
* Considered by the investigator to have poor compliance.
* Any other significant disease or condition that, in the investigator's judgment, may jeopardize the subject's safety or interfere with the study assessments.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events as Assessed by CTCAE V5.0 | 52 weeks post-transplant
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs).

SECONDARY OUTCOMES:
Change from baseline in the UMSARS total score (Part I + Part II) at Weeks 13, 26, and 52. | Weeks 13, 26, and 52 post-transplant
  Change from baseline in the Unified Multiple System Atrophy Rating Scale (UMSARS) total score (Part I Score 0 ~ 48 + Part II Score 0 ~ 56; ) at Weeks 13, 26, and 52. A higher score indicates more severe symptoms or worse health.
Change from baseline in the UMSARS Part I score at Weeks 13, 26, and 52. | Weeks 13, 26, and 52 post-transplant
  Change from baseline in the Unified Multiple System Atrophy Rating Scale (UMSARS) Part I score (0 ~ 48) at Weeks 13, 26, and 52. A higher score indicates more severe symptoms or worse health.
Change from baseline in the UMSARS Part II score at Weeks 13, 26, and 52. | Weeks 13, 26, and 52 post-transplant
  Change from baseline in the Unified Multiple System Atrophy Rating Scale (UMSARS) Part II score (0 ~ 56) at Weeks 13, 26, and 52. A higher score indicates more severe symptoms or worse health.
Change from baseline in dopaminergic metabolism of the basal ganglia at Week 52, as measured by DAT PET imaging. | Weeks 52 post-transplant
  Change from baseline in dopaminergic metabolism of the basal ganglia at Week 52, as measured by 18F-DOPA PET or 11C-CFT DAT PET imaging.
Change from baseline in the CGI-S score at Weeks 13, 26, and 52. | Weeks 13, 26, and 52 post-transplant
  Change from baseline in the Clinical Global Impression-Severity scale (CGI-S) score (1 ~ 7) at Weeks 13, 26, and 52. A higher score indicates more severe symptoms or worse health.

OTHER OUTCOMES:
Pharmacodynamic Biomarkers (NfL) | Weeks 13, 26, and 52 post-transplant
  measurement of neurofilament light chain (NfL) levels in human blood samples.
Pharmacodynamic Biomarkers (α-syn) | Weeks 13, 26, and 52 post-transplant
  measurement of alpha-synuclein (α-syn) levels in human blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China